CLINICAL TRIAL: NCT03453983
Title: Transcranial Direct Current Stimulation (tDCS): A Therapeutic Intervention for Motor Impairments in Children With Developmental Coordination Disorder (DCD).
Brief Title: Does tDCS Improve Motor Learning in Children With DCD?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB18-0183
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2019-04

CONDITIONS: Developmental Coordination Disorder
Keywords: Neurodevelopment; Pediatrics; Motor Learning; Brain Imaging; Neuroscience
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Intervention Model Description: The currently proposed study is a randomized, sham controlled clinical trial that includes 30 adolescents diagnosed with DCD. Participants will be randomized to one of two tDCS treatment groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be informed of the stimulation group to which they are randomized. Both stimulation groups produce similar transient scalp sensations in participants and the sham protocol that will be used has been shown to be valid and ensures that participants are naïve to their assigned treatment group [9]. Participants will be asked which stimulation group they felt they took part in to ensure adequate blinding.
  Outcomes assessors will be blinded. Offline video analysis will be used to score motor assessment performance. These videos will exclude all identifying information including the participant's face and their stimulation group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal tDCS Intervention Group (Experimental): Transcrainial Direct Current Stimulation (tDCS): The right primary motor cortex will be localized and a saline soaked sponge electrode will be placed onto M1 with a second saline soaked sponge electrode placed on the contralateral supraorbital region.
  Interventions: Device: Transcrainial Direct Current Stimulation (tDCS)
- Sham tDCS Intervention Group (Sham Comparator): Transcrainial Direct Current Stimulation (tDCS): The right primary motor cortex will be localized and a saline soaked sponge electrode will be placed onto M1 with a second saline soaked sponge electrode placed on the contralateral supraorbital region.
  Interventions: Device: Transcrainial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcrainial Direct Current Stimulation (tDCS) — Transcranial direct current stimulation (tDCS) is a safe non-invasive form of brain stimulation, which modulates, through the application of weak direct current, cortical excitability. The applied subthreshold current passes through two externally placed electrodes, an anode and cathode.

SUMMARY:
Transcrainial direct current stimulation (tDCS) has become increasingly popular over the past decade. tDCS is a safe and well-studied form of non-invasive brain stimulation. The purpose of the current study is to see if tDCS can improve motor function in children with developmental coordination disorder.

Non-invasive brain stimulation is shown to positively affect motor performance in children with neurodevelopmental and/or neurological conditions. For example, tDCS improves hand motor function in children with paediatric stroke and cerebral palsy. The benefits of tDCS in developmental coordination disorder is unknown. The current study will assess children's motor performance before and after tDCS intervention.

DETAILED DESCRIPTION:
Developmental Coordination Disorder (DCD) is a chronic neurodevelopmental disorder characterized by impairments in coordinated motor abilities. Affected individuals show differences in brain maturation and early motor development, negatively impacting performance on everyday living tasks such as writing and participation in sports. Currently, there are few evidence-based therapeutic interventions for individuals diagnosed with DCD, and most are time consuming with modest effect sizes [1]. There is a pressing need to develop efficient, effective interventions to improve motor performance in children with DCD, as impairments often last into adulthood and can negatively impact long-term physical and mental health as well as social and academic abilities.

The ability to enhance endogenous motor learning systems with non-invasive brain stimulation is now well established in adults [2, 3]. Research studies have demonstrated the same potential in the developing brain. For instance, tDCS can significantly enhance the acquisition of motor skills over a few brief training sessions in typically developing school aged children, with lasting effects [4]. Recent clinical trials in children with cerebral palsy and neonatal stroke also suggest therapeutic efficacy in children with motor impairment [5, 6, 7]. However, the use of tDCS in pediatric populations is limited [8]. As tDCS has been associated with improved motor outcomes in adults and children with motor impairment, it may be an effective intervention for children with DCD. This however has not been investigated.

Research Questions & Objectives:

The current study will investigate the therapeutic benefits of tDCS in adolescents with DCD. The primary aim is to determine changes in motor skill acquisition and learning during a skill-training paradigm that is paired with anodal tDCS or sham tDCS. We hypothesize that when compared to the sham tDCS group, the treatment tDCS group will show enhanced motor learning on tests of motor functioning.

Secondarily we will also examine sensorimotor changes following tDCS intervention and pediatric brain stimulation safety/tolerability.

Methods:

A randomized, sham controlled clinical trial including a final sample of 30 school aged children diagnosed with DCD will be conducted. The current study will be using a well-supported stimulation protocol, utilized in children and adolescents in the absence of adverse side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed and documented DCD (including individuals with additional diagnoses of attention and/or learning disorders)
* Aged 10 to 15 years
* Right Handed

Exclusion Criteria:

* Presence of implanted electrical devices, metallic implants, and/or irremovable metal objects (i.e., cardiac pacemakers, braces etc.)
* Pregnancy or possibility of pregnancy
* Diagnosed with a neuropsychiatric disorder such as autism spectrum disorder or chronic medical condition such as cerebral palsy or epilepsy
* Taking prescribed medications

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Purdue Pegborad Test (PPT) | 20 minutes
  The PPT is a valid measure of fine motor coordination, hand dexterity, and motor learning skills, which consists of 4 subtests: left hand peg placement [PPTL], right hand peg placement [PPTR], bimanual peg placement [PPTLR], and bimanual assembly [PPTA]. The PPT peg placement subtests involve placing as many pins as possible into a pegboard during a 30 second interval. The total number of pegs, or pairs of pegs, placed are counted and scored. The PPT assembly subtest involved building as many copies of a demonstration structure using pins, pegs, and washers within a 60 second time period.

SECONDARY OUTCOMES:
Jebsen-Taylor Test of Hand Function (JTT) | 20 minutes
  The JTT is an upper extremity motor assessment aimed at testing practical everyday living skills, such as writing, picking up coins, and moving objects. Left and right hands are tested independently, and scores for each hand are obtained through recording task completion time.
Serial Reaction Time Task (SRTT) | 20 minutes
  The SRTT is a measure of motor learning skills. Participants are cued on a computer monitor to press the indicated letter on the keyboard. Participants complete this task over eight blocks of trials, each consisting of 96 cued key commands.

OTHER OUTCOMES:
KINARM | 45 minutes
  Sensorimotor changes will be measured between baseline, post-training, and 6 week follow-up using the Kinesiological Instrument for Normal and Altered Reaching Movements (KINARM, BKIN Technologies Ltd, Ontario, Canada). The KINARM robot is a valid and reliable tool that can be used to measure children's proprioceptive, sensorimotor, visuomotor and motor decision/control abilities.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah M Dewey, PhD, Principal Investigator — University of Calgary
Locations (1):
- Child Development Center, Owerko Centre Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Currently, there is no pre-determined plan to share any collected data with other researchers.

REFERENCES:
- [Background] Smits-Engelsman BC, Blank R, van der Kaay AC, Mosterd-van der Meijs R, Vlugt-van den Brand E, Polatajko HJ, Wilson PH. Efficacy of interventions to improve motor performance in children with developmental coordination disorder: a combined systematic review and meta-analysis. Dev Med Child Neurol. 2013 Mar;55(3):229-37. doi: 10.1111/dmcn.12008. Epub 2012 Oct 29. PMID 23106530
- [Background] Reis J, Schambra HM, Cohen LG, Buch ER, Fritsch B, Zarahn E, Celnik PA, Krakauer JW. Noninvasive cortical stimulation enhances motor skill acquisition over multiple days through an effect on consolidation. Proc Natl Acad Sci U S A. 2009 Feb 3;106(5):1590-5. doi: 10.1073/pnas.0805413106. Epub 2009 Jan 21. PMID 19164589
- [Background] Goodwill AM, Reynolds J, Daly RM, Kidgell DJ. Formation of cortical plasticity in older adults following tDCS and motor training. Front Aging Neurosci. 2013 Dec 6;5:87. doi: 10.3389/fnagi.2013.00087. eCollection 2013. PMID 24367333
- [Background] Ciechanski P, Kirton A. Transcranial Direct-Current Stimulation Can Enhance Motor Learning in Children. Cereb Cortex. 2017 May 1;27(5):2758-2767. doi: 10.1093/cercor/bhw114. PMID 27166171
- [Background] Kirton A, Ciechanski P, Zewdie E, Andersen J, Nettel-Aguirre A, Carlson H, Carsolio L, Herrero M, Quigley J, Mineyko A, Hodge J, Hill M. Transcranial direct current stimulation for children with perinatal stroke and hemiparesis. Neurology. 2017 Jan 17;88(3):259-267. doi: 10.1212/WNL.0000000000003518. Epub 2016 Dec 7. PMID 27927938
- [Background] Kirton A, Andersen J, Herrero M, Nettel-Aguirre A, Carsolio L, Damji O, Keess J, Mineyko A, Hodge J, Hill MD. Brain stimulation and constraint for perinatal stroke hemiparesis: The PLASTIC CHAMPS Trial. Neurology. 2016 May 3;86(18):1659-67. doi: 10.1212/WNL.0000000000002646. Epub 2016 Mar 30. PMID 27029628
- [Background] Moura RCF, Santos C, Collange Grecco L, Albertini G, Cimolin V, Galli M, Oliveira C. Effects of a single session of transcranial direct current stimulation on upper limb movements in children with cerebral palsy: A randomized, sham-controlled study. Dev Neurorehabil. 2017 Aug;20(6):368-375. doi: 10.1080/17518423.2017.1282050. Epub 2017 Feb 25. PMID 28632467
- [Background] Bikson M, Grossman P, Thomas C, Zannou AL, Jiang J, Adnan T, Mourdoukoutas AP, Kronberg G, Truong D, Boggio P, Brunoni AR, Charvet L, Fregni F, Fritsch B, Gillick B, Hamilton RH, Hampstead BM, Jankord R, Kirton A, Knotkova H, Liebetanz D, Liu A, Loo C, Nitsche MA, Reis J, Richardson JD, Rotenberg A, Turkeltaub PE, Woods AJ. Safety of Transcranial Direct Current Stimulation: Evidence Based Update 2016. Brain Stimul. 2016 Sep-Oct;9(5):641-661. doi: 10.1016/j.brs.2016.06.004. Epub 2016 Jun 15. PMID 27372845
- [Background] Ambrus GG, Al-Moyed H, Chaieb L, Sarp L, Antal A, Paulus W. The fade-in--short stimulation--fade out approach to sham tDCS--reliable at 1 mA for naive and experienced subjects, but not investigators. Brain Stimul. 2012 Oct;5(4):499-504. doi: 10.1016/j.brs.2011.12.001. Epub 2012 Feb 22. PMID 22405745
- [Derived] Grohs MN, Craig BT, Kirton A, Dewey D. Effects of Transcranial Direct Current Stimulation on Motor Function in Children 8-12 Years With Developmental Coordination Disorder: A Randomized Controlled Trial. Front Hum Neurosci. 2020 Dec 11;14:608131. doi: 10.3389/fnhum.2020.608131. eCollection 2020. PMID 33362497